CLINICAL TRIAL: NCT06603506
Title: Collection of Endometrial Cancer-derived Organoids to Evaluate the Efficacy of PARP Inhibitors: PENDOR Pilot Study
Acronym: PENDOR
Status: Recruiting | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A01206-41; 2024-A01206-41 (Other: ID-RCB number)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; organoide; PARP inhibitor
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- tumour and blood collection: tumour and blood collection for realization ex vivo organoid models
  Interventions: Other: tumour and blood samples

INTERVENTIONS:
Other: tumour and blood samples — Tumour and blood samples

SUMMARY:
This study comprises 3 stages:

1. Collection of tumor and blood samples.
2. Creation of organoid models based on tumor samples.
3. Development of functional tests to predict clinical response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or more
* Patient with histologically confirmed, localized endometrial cancer, candidate for surgical treatment.
* Patient with localized endometrial cancer, presenting:

  * A high-grade endometrioid histological type and/or
  * P53 mutation and/or
  * a non-endometrioid histological type regardless of P53 status.
* Patient affiliated to a social security scheme
* Information and signature of informed consent prior to any specific study procedure

Exclusion Criteria:

* Other active cancer less than 6 months old (with the exception of treated basal cell carcinoma of the skin).
* Patient deprived of liberty, under guardianship, or subject to a legal protection measure, or unable to express consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with localized endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Rate of establishment of exploitable tumor organoid lines | through study completion, an average of 3 years
  Rate of establishment of tumor organoid lines usable for predictive assays of response to PARP inhibitors.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gall GL, Cherifi F, Divoux J, Florent R, Christy F, Leconte A, San C, Devillers A, Desmartin G, Lecouflet L, Clarisse B, Ballesta S, Thorel L, Dubois B, Harter V, Rousseau N, Gaichies L, Martin-Francoise S, Le Brun JF, Dolivet E, Rouzier R, Jeanne C, Blanc-Fournier C, Figeac M, Leman R, Castera L, Poulain L, Weiswald LB, Joly F. The PENDOR study: establishment of a panel of patient-derived tumor organoids from endometrial cancer to assess efficacy of PARP inhibitors. BMC Cancer. 2025 Feb 11;25(1):244. doi: 10.1186/s12885-025-13590-6. PMID 39934735